CLINICAL TRIAL: NCT04175028
Title: Neuromodulation of Executive Function in the ADHD Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2014P001401
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Executive Function
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ADHD (Other): Patients with ADHD.
  Interventions: Device: Transcranial Direct Current Stimulation
- Healthy Control (Other): Volunteers without Neuropsychiatric Disorders.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, electrodes are applied on the scalp to transmit direct current at low current amplitudes.

SUMMARY:
This study aims to determine the transient, modulatory effects of transcranial direct current stimulation (tDCS) on executive function and inhibitory control in patients with ADHD compared to healthy controls.

DETAILED DESCRIPTION:
This study aims to determine the transient, modulatory effects of transcranial direct current stimulation (tDCS) on executive function and inhibitory control in patients with ADHD. Deficits in these cognitive functions are core to ADHD, and cause significant impairment and morbidity. The study will also include a cohort of healthy controls for comparison.

ELIGIBILITY:
Inclusion Criteria

1. Male and female subjects 18-66 years of age
2. Healthy volunteers or volunteers with a diagnosis of ADHD in adulthood, meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) [American Psychiatric Association, 2013] criteria, including at least 5 moderate inattentive or impulsive-hyperactive symptoms, and onset of two symptoms of inattentive or of impulsive/hyperactive traits by the age of 12.
3. Patient will be either off stimulant medications or, if undergoing treatment with stimulants, will be asked to discontinue two days prior to the experiment, under physician-guided protocol, and allowed to resume afterwards. Subjects may resume stimulant use between the two study visits so long as they discontinue use two days prior to the second study visit. If fatigue is problematic in subjects discontinuing medication, they will be allowed to continue with the study if they are able to follow the suggested taper plan (50% of the dose day one, 25% dose day 2, stop day of visit (day 3)).
4. English-speaking

Exclusion Criteria

1. Current or past history of clinically unstable psychiatric conditions such as suicidal or homicidal behavior or psychotic disorders.
2. Pregnant or nursing females.
3. Inability to participate in testing procedures
4. Contraindication to tDCS: history or epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, VP shunt, pacemakers, pregnancy.
5. Additional exclusion criteria for healthy controls:

   1. Diagnosis of psychiatric of neurological disorder
   2. Ongoing treatment with any psychotropic medications.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Accuracy and Reaction Time in Attention and Working Memory | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  N-Back Task
Change in Accuracy and Reaction Time in Attention and Working Memory | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  Flanker Task
Change in Accuracy and Reaction Time in Attention and Working Memory | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  Multi-Source Interference with International Affective Picture System Task
Change in Accuracy and Reaction Time in Inhibition/Decision Making | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  Delayed Discounting
Change in Accuracy and Reaction Time in Inhibition/Decision Making | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  Stop Signal Task
Change in Accuracy and Reaction Time in Inhibition/Decision Making | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  Cambridge Gambling Task

SECONDARY OUTCOMES:
Amplitude of Encephalogram (EEG) Event Related Potentials | Change Before and After Stimulation on Each of the Three Visits, Average 2-6 Weeks
  Measure of amplitude related to stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PhD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubreuil-Vall L, Gomez-Bernal F, Villegas AC, Cirillo P, Surman C, Ruffini G, Widge AS, Camprodon JA. Transcranial Direct Current Stimulation to the Left Dorsolateral Prefrontal Cortex Improves Cognitive Control in Patients With Attention-Deficit/Hyperactivity Disorder: A Randomized Behavioral and Neurophysiological Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Apr;6(4):439-448. doi: 10.1016/j.bpsc.2020.11.006. Epub 2020 Nov 25. PMID 33549516